CLINICAL TRIAL: NCT01335451
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD5213 After Oral Administration of Single and Multiple Ascending Doses in Healthy Young and Elderly J
Brief Title: Assess the Safety, Tolerability and Pharmacokinetics of AZD5213 After Single and Multiple Ascending Oral Doses in Healthy Young and Elderly Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D3030C00004
Record Dates: First submitted 2011-04-13; First posted 2011-04-14 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: AZD5213; safety; pharmacokinetics; single dose; repeated dose; young; elderly; Japanese; healthy subject

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Each cohort will have 6 subjects that will receive AZD5213
  Interventions: Drug: AZD5213
- Placebo (Placebo Comparator): Each cohort will have 2 subjects that will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5213 — Four increasing doses for young and two increasing doses for elderly subjects. Subject will receive single dose of AZD5213 oral solution (Day 1) and then start the once daily repeated doses from Day 3 to 12 for 10 days
  Arms: Active
Drug: Placebo — Placebo solution, single dose (Day 1) and repeated dose from Day 3 to 12 for 10 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety, tolerability and pharmacokinetics of AZD5213 in healthy young and elderly Japanese subjects

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Japanese healthy male subjects aged 20 to 45 years (young) and male and female subjects aged 65 to 80 years (elderly)
* Male subjects should be willing to use barrier contraception ie, condoms, from the first day of dosing until 3 months after the last dose of investigational product
* Have a body mass index (BMI) between 17 and 27 kg/m2 and weigh at least 45 kg and no more than 100 kg
* Clinically normal physical findings, supine BP, pulse rate, ECG and laboratory assessments in relation to age, as judged by the investigator(s)

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* History of previous or ongoing psychiatric disease/condition including psychosis, affective disorder, anxiety disorder, and personality disorder including borderline according to the criteria in the Diagnostic and Statistical Manual of Mental Disorders
* History of psychotic disorder among first degree relatives.
* History of use of antipsychotic, antidepressant or anxiolytic drugs, prescribed as well as non-prescribed use.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of AZD5213 by assessment of adverse event, vital signs, laboratory parameters and electrocardiograms (ECGs). | Range of Days 1-12

SECONDARY OUTCOMES:
To assess the PK of AZD5213 after a single and multiple doses by assessment of Cmax. | Range of Days 1-12
To assess the PK of AZD5213 after a single and multiple doses by assessment of fe. | Range of Days 1-12
To assess the PK of AZD5213 after a single and multiple doses by assessment of CLR. | Range of Days 1-12
To assess the PK of AZD5213 after a single and multiple doses by assessment of CL/F. | Range of Days 1-12
To assess the PK of AZD5213 after a single and multiple doses by assessment of t1/2. | Range of Days 1-12
To assess the PK of AZD5213 after a single and multiple doses by assessment of tmax. | Range of Days 1-12
To assess the PK of AZD5213 after a single and multiple doses by assessment of AUC. | Range of Days 1-12

CONTACTS AND LOCATIONS:
Overall Officials: Märta Segerdahl, MD, PhD, Study Director — AstraZeneca R&D, Södertälje; Akimasa Watanabe, MD, Principal Investigator — Kyushu Clinical Pharmacology Research Clinic, Japan
Locations (1):
- Research Centre, Fukuoka, Japan

REFERENCES:
- See also: D3030C00004_Clinical_Study_Report_Synopsis.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1315&filename=D3030C00004_Clinical_Study_Report_Synopsis.pdf